CLINICAL TRIAL: NCT06422520
Title: A Phase 1 Study Investigating the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of BGB-C354, an Antibody-Drug Conjugate Targeting B7H3, Alone and in Combination With Anti-PD-1 Monoclonal Antibody Tislelizumab in Patients With Advanced Solid Tumors
Brief Title: A First-in-Human Study of BGB-C354 Alone and in Combination With Tislelizumab in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-C354-101; 2024-513280-11-00 (EU CTIS Number)
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor
Keywords: BGB-C354; Tislelizumab; First-in-human; Advanced solid tumor; Anti-PD-1 Monoclonal Antibody; B7H3; antibody drug conjugate
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1a: Part A (Monotherapy Dose Escalation) (Experimental): BGB-C354 monotherapy doses at sequentially increasing levels.
  Interventions: Drug: BGB-C354
- Phase 1a: Part B (Safety Expansion) (Experimental): Participants will enroll at safe dose levels recommended by the Safety Monitoring Committee (SMC) for further evaluation.
  Interventions: Drug: BGB-C354
- Phase 1b: Part C (Monotherapy Expansion) (Experimental): BGB-C354 will be administered at the recommended dose for expansion (RDFE).
  Interventions: Drug: BGB-C354
- Phase 1b: Part D (Combination Therapy Expansion) (Experimental): BGB-C354 and tislelizumab will be adminsitered at doses determined by the SMC.
  Interventions: Drug: BGB-C354; Drug: Tislelizumab

INTERVENTIONS:
Drug: BGB-C354 — Administered by intravenous infusion
Drug: Tislelizumab — Administered by intravenous infusion
  Arms: Phase 1b: Part D (Combination Therapy Expansion)

SUMMARY:
This is a first-in-human, Phase 1a/1b study to evaluate the safety, tolerability, pharmacokinetics, and preliminary antitumor activity of BGB-C354 alone and in combination with tislelizumab in participants with advanced solid tumors.

Study details include:

* The study will be conducted in 2 phases: Phase 1a (Monotherapy Dose Escalation and Safety Expansion) and Phase 1b (Dose Expansion).
* The visit frequency will be approximately every 21 days during study treatment. Maximum treatment duration will be up to two years.
* The study duration is estimated to be approximately 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide a signed and dated written informed consent prior to any study-specific procedures, sampling, or data collection.
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
3. Participants with histologically or cytologically confirmed advanced, metastatic, or unresectable solid tumors, whose cancer is not amenable to therapy with curative intent:
4. ≥ 1 measurable lesion per RECIST v1.1.
5. Able to provide an archived tumor tissue sample.
6. Adequate organ function.
7. Females of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study, and for ≥ 7 months after the last dose of study drug(s).
8. Nonsterile males must be willing to use a highly effective method of birth control for the duration of the study treatment period and for ≥ 4 months after the last dose of study drug(s).

Exclusion Criteria:

1. Prior treatment with B7H3-targeted therapy.
2. For Part B and Phase 1b: Prior treatment with antibody drug conjugates (ADCs) with topoisomerase I inhibitor payload (for Phase 1b, unless otherwise specified for specific cohorts).
3. Participants with spinal cord compressions, active leptomeningeal disease or uncontrolled, or untreated brain metastasis
4. Any malignancy ≤ 2 years before the first dose of study treatment(s) except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated with curative intent (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast).
5. History of interstitial lung disease, ≥ Grade 2 noninfectious pneumonitis, oxygen saturation at rest < 92%, or requirement for supplemental oxygen at baseline
6. Uncontrolled diabetes, or > Grade 1 laboratory test abnormalities in potassium, sodium, or corrected calcium levels despite standard medical management ≤ 14 days before the first dose of study drug(s).
7. Infection (including tuberculosis infection) requiring systemic (oral or intravenous) antibacterial, antifungal, or antiviral therapy ≤ 14 days before the first dose of study treatment(s).

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Approximately 24 months
  Number of participants with AEs and SAEs characterized by type, frequency, severity (as graded by the National Cancer Institute- Common Terminology Criteria for Adverse Events Version 5.0 [NCI-CTCAE v 5.0]), timing, seriousness, and relationship to study drug(s); physical examinations; electrocardiograms (ECGs); and laboratory assessments as needed; and adverse events meeting protocol-defined dose-limiting toxicity (DLT) criteria
Phase 1a: Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) of BGB-C354 | Approximately 1 month
  Defined as the highest dose evaluated for which the estimated toxicity rate is closest to the target toxicity rate of 30% or the highest dose administered, respectively
Phase 1a: Recommended Dose for Expansion (RDFE) of BGB-C354 | Approximately 24 months
  The potential RDFE(s) of BGB-C354 will be determined based on the MTD or MAD, taking into consideration the long-term tolerability, pharmacokinetics (PK), preliminary antitumor activity, and any other relevant data, as available
Phase 1b: Overall Response Rate (ORR) | Approximately 24 months
  ORR is defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR) assessed by the investigator using Response Evaluations Criteria in Solid Tumors Version 1.1 (RECIST v1.1).
Phase 1b: Recommended Phase 2 dose (RP2D) of BGB-C354 alone and in combination with tislelizumab | Approximately 24 months
  The RP2D of BGB-C354 will be determined based on safety, PK, pharmacodynamics, preliminary antitumor activity, and other relevant data, as available.

SECONDARY OUTCOMES:
Phase 1a: ORR | Approximately 24 months
  ORR is defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR) assessed by the investigator using RECIST v1.1.
Duration of Response (DOR) | Approximately 24 months
  DOR is defined as the time from the first determination of an objective response per RECIST v1.1 until the first documentation of disease progression or death, whichever occurs first as assessed by the investigator.
Disease Control Rate (DCR) | Approximately 24 months
  DCR is defined as the percentage of participants with best overall response of CR, PR, or stable disease as determined from tumor assessments by the investigator using RECIST v1.1.
Phase 1b: Progression Free Survival (PFS) | Approximately 24 months
  PFS is defined as the time from the date of the first dose of study drug(s) to the date of the first documentation of progressive disease assessed by the investigator using RECIST v1.1 or death, whichever occurs first as determined from tumor assessments by the investigator using RECIST v1.1.
Phase 1b: Number of Participants with Adverse Events (AEs) and Serious Adverse Events | Approximately 24 months
  Number of participants with AEs and SAEs characterized by type, frequency, severity (as graded by the National Cancer Institute- Common Terminology Criteria for Adverse Events Version 5.0 [NCI-CTCAE v 5.0]), timing, seriousness, and relationship to study drug(s); physical examinations; electrocardiograms (ECGs); and laboratory assessments as needed; and adverse events meeting protocol-defined dose-limitingtoxicity (DLT) criteria
Maximum observed plasma concentration (Cmax) for BGB-C354 | Twice in the first 3 months
Minimum observed plasma concentration (Cmin) for BGB-C354 | Approximately 12 months
Time to maximum plasma concentration (Tmax) for BGB-C354 | Twice in the first 3 months
Half-life (t1/2) for BGB-C354 | Twice in the first 3 months
Area under the concentration-time curve (AUC) for BGB-C354 | Twice in the first 3 months
Apparent clearance (CL/F) for BGB-C354 | Approximately 12 months
Apparent volume of distribution (Vz/F) for BGB-C354 | Approximately 12 months
Accumulation ratio for BGB-C354 | Approximately 12 months
Number of participants with anti-drug antibodies (ADAs) to BGB-C354 | Approximately 12 months
Serum concentration of BGB-C354 | Approximately 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (14):
- United States (5):
  - Florida Cancer Specialist Research Institute Lake Nona, Orlando, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Next Oncology, Austin, Texas
  - The University of Texas Md Anderson Cancer Center, Houston, Texas
- Australia (4):
  - Westmead Hospital, Westmead, New South Wales
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - One Clinical Research, Nedlands, Western Australia
- China (5):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Jilin Cancer Hospital, Changchun, Jilin
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/